CLINICAL TRIAL: NCT02980887
Title: Redefining Pulmonary Hypertension Through Pulmonary Vascular Disease Phenomics (PVDOMICS)
Brief Title: Pulmonary Vascular Disease Phenomics Program PVDOMICS
Acronym: PVDOMICS
Status: Active, not recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Brigham and Women's Hospital (Other); Columbia University (Other); Weill Medical College of Cornell University (Other); Johns Hopkins University (Other); Mayo Clinic (Other); University of Arizona (Other); Vanderbilt University (Other)
Responsible Party: Sponsor
Other Study IDs: 16-860
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary arterial hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples for Omics analyses, including DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Controls: Healthy controls No intervention as this is an observational study
  Interventions: Other: No Intervention
- Pulmonary Vascular Disease: Pulmonary Vascular Disease at risk for pulmonary hypertension
  Interventions: Other: No Intervention
- Pulmonary Hypertension: Those meeting WSPH/WHO group classifications 1-5 of pulmonary hypertension
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — There is no intervention in this observational study

SUMMARY:
It is recognized that patients with various forms of heart and lung disease exhibit varying degrees of pulmonary hypertension, pulmonary vascular remodeling, and right ventricular dysfunction. The genetic, molecular, and cellular processes driving these phenomena are not well understood. Rapid advances in high throughput omic methodology, combined with powerful bioinformatics and network biology capability, have created the opportunity to conduct studies that broadly search for homologies and differences across the spectrum of disease states associated with pulmonary hypertension, and determinants of the spectrum of right ventricular compensation that accompanies these conditions

DETAILED DESCRIPTION:
The protocol is designed to lead to new understanding of patients with pulmonary hypertension and right heart dysfunction, based on molecular, clinical, hemodynamic and radiographic characteristics. New classifications will be a product of association of these in depth phenotypic descriptions with specific molecular mechanisms of pathogenesis. The protocol will be implemented to lead to identification of both sub-phenotypes of lung vascular disease and to biomarkers of disease that may be useful for early diagnosis or for assessment of interventions to prevent or treat this condition.

A longitudinal study in a subset of the participants enrolled in the parent cross-sectional study will:

1. Retest participants at a minimum 6 month interval from initial evaluation to collect a core set of clinical and OMICS features. This will include survival, clinical staging, clinical group assignment, 6-minute walk, echocardiography, and blood for a broad collection of selected OMICS tests, to include proteomics and other variables found to be informative in the initial set.
2. Associate and compare OMICS data with clinical sets and OMICS clusters between baseline and follow-up interval, with attention to reproducibility, predictive capacity as biomarkers for diagnosis, disease progression, phenotypic changes, functional capacity, therapeutic response and survival.

ELIGIBILITY:
Cross-sectional (parent) study:

Inclusion Criteria:

Patients ages >18 years of age referred for right heart catheterization for further evaluation of known PVD or to be at risk for PVD due to established cardiac disease or pulmonary disease

* Able to perform complete diagnostic testing listed subsequently (cardiac catheterization, echo, exercise test, PFT's, ECG, chest CT, quality of life questionnaires, ventilation/perfusion scan, cardiac MRI, body composition bioimpedance, and sleep study)
* Subject signs informed consent to perform required testing for the protocol

Exclusion Criteria:

Dialysis dependent renal function; In the clinician's opinion, too ill to perform the protocol testing; Pregnant or nursing

Longitudinal study:

Inclusion Criteria:

* Any PH, comparators or control participant previously enrolled in the parent PVDOMICS protocol with a minimum of six months post-enrollment
* Dialysis dependent renal function since the parent study acceptable

Exclusion Criteria:

Participant Level 1 (clinic visit):

* Transplant other than heart or lung
* In the clinician's opinion, too ill to perform L-PVDOMICS testing even if limited testing.
* Participants who withdrew from the parent PVDOMICS study
* Pregnant or nursing
* Concurrent participation in any investigational drug study or other clinical trial

Participant Level 2 (telephone visit):

* Transplant other than heart or lung
* Participants who withdrew from the parent PVDOMICS study

Participant Level 3 (medical chart review):

- Participants who withdrew from the parent PVDOMICS study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary hypertension, Pulmonary hypertension vascular, and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 1195 (Actual)
Dates: Start 2016-11; Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Precision based definitions of pulmonary vascular diseases (PVD) | Over 5 years
  OMICs analyses will be used to assign new class of PVD

SECONDARY OUTCOMES:
Identification of biomarkers for PVD | 5 years
  OMICs and other measures of disease

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S Hill, MD, Study Chair — Tufts University Medical Center; Lei Xiao, MD, Study Director — National Heart, Lung, and Blood Institute (NHLBI)
Locations (7):
- United States (7):
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Weill Cornell Medicine, New York, New York
  - New York Medical College, Valhalla, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Plan for sharing with outside network investigators is being developed. Data will be archived at BioLINCC and BioDataCatalyst.
Supporting Information: Study Protocol, ICF
Time Frame: Being determined
Access Criteria: Being decided

REFERENCES:
- [Background] Hemnes AR, Leopold JA, Radeva MK, Beck GJ, Abidov A, Aldred MA, Barnard J, Rosenzweig EB, Borlaug BA, Chung WK, Comhair SAA, Desai AA, Dubrock HM, Erzurum SC, Finet JE, Frantz RP, Garcia JGN, Geraci MW, Gray MP, Grunig G, Hassoun PM, Highland KB, Hill NS, Hu B, Kwon DH, Jacob MS, Jellis CL, Larive AB, Lempel JK, Maron BA, Mathai SC, McCarthy K, Mehra R, Nawabit R, Newman JH, Olman MA, Park MM, Ramos JA, Renapurkar RD, Rischard FP, Sherer SG, Tang WHW, Thomas JD, Vanderpool RR, Waxman AB, Wilcox JD, Yuan JX, Horn EM; PVDOMICS Study Group. Clinical Characteristics and Transplant-Free Survival Across the Spectrum of Pulmonary Vascular Disease. J Am Coll Cardiol. 2022 Aug 16;80(7):697-718. doi: 10.1016/j.jacc.2022.05.038. PMID 35953136
- [Background] Hemnes AR, Beck GJ, Newman JH, Abidov A, Aldred MA, Barnard J, Berman Rosenzweig E, Borlaug BA, Chung WK, Comhair SAA, Erzurum SC, Frantz RP, Gray MP, Grunig G, Hassoun PM, Hill NS, Horn EM, Hu B, Lempel JK, Maron BA, Mathai SC, Olman MA, Rischard FP, Systrom DM, Tang WHW, Waxman AB, Xiao L, Yuan JX, Leopold JA; PVDOMICS Study Group. PVDOMICS: A Multi-Center Study to Improve Understanding of Pulmonary Vascular Disease Through Phenomics. Circ Res. 2017 Oct 27;121(10):1136-1139. doi: 10.1161/CIRCRESAHA.117.311737. PMID 29074534
- [Derived] Menon DP, Frantz RP, Gochanour BR, Beck GJ, Berman-Rosenzweig ES, Borlaug BA, Erzurum SC, Farha S, Finet JE, Grunig G, Hassoun PM, Hemnes AR, Hill NS, Horn EM, Lempel JK, Leopold JA, Mathai SC, Renapurkar RD, Rischard FP, Waxman AB, DuBrock HM. Ground-Glass Opacities in Pulmonary Arterial Hypertension-Results from the PVDOMICS Study. Ann Am Thorac Soc. 2025 Dec;22(12):1863-1873. doi: 10.1513/AnnalsATS.202503-333OC. PMID 40680159
- [Derived] Reddy YNV, Frantz RP, Hemnes AR, Hassoun PM, Horn E, Leopold JA, Rischard F, Rosenzweig EB, Hill NS, Erzurum SC, Beck GJ, Finet JE, Jellis CL, Mathai SC, Tang WHW, Borlaug BA; PVDOMICS Study Group. Disentangling the Impact of Adiposity From Insulin Resistance in Heart Failure With Preserved Ejection Fraction. J Am Coll Cardiol. 2025 May 13;85(18):1774-1788. doi: 10.1016/j.jacc.2025.03.530. PMID 40335254
- [Derived] Borlaug BA, Larive B, Frantz RP, Hassoun P, Hemnes A, Horn E, Leopold J, Rischard F, Berman-Rosenzweig E, Beck G, Erzurum S, Farha S, Finet JE, Highland KB, Jacob M, Jellis C, Mehra R, Renapurkar R, Singh H, Tang WHW, Vanderpool R, Wilcox J, Yu S, Hill N. Pulmonary hypertension across the spectrum of left heart and lung disease. Eur J Heart Fail. 2024 Jul;26(7):1642-1651. doi: 10.1002/ejhf.3302. Epub 2024 Jun 4. PMID 38837273
- [Derived] Lowery MM, Hill NS, Wang L, Rosenzweig EB, Bhat A, Erzurum S, Finet JE, Jellis CL, Kaur S, Kwon DH, Nawabit R, Radeva M, Beck GJ, Frantz RP, Hassoun PM, Hemnes AR, Horn EM, Leopold JA, Rischard FP, Mehra R; Pulmonary Vascular Disease Phenomics (PVDOMICS) Study Group. Sleep-Related Hypoxia, Right Ventricular Dysfunction, and Survival in Patients With Group 1 Pulmonary Arterial Hypertension. J Am Coll Cardiol. 2023 Nov 21;82(21):1989-2005. doi: 10.1016/j.jacc.2023.09.806. PMID 37968017
- [Derived] Tang WHW, Wilcox JD, Jacob MS, Rosenzweig EB, Borlaug BA, Frantz RP, Hassoun PM, Hemnes AR, Hill NS, Horn EM, Singh HS, Systrom DM, Tedford RJ, Vanderpool RR, Waxman AB, Xiao L, Leopold JA, Rischard FP. Comprehensive Diagnostic Evaluation of Cardiovascular Physiology in Patients With Pulmonary Vascular Disease: Insights From the PVDOMICS Program. Circ Heart Fail. 2020 Mar;13(3):e006363. doi: 10.1161/CIRCHEARTFAILURE.119.006363. Epub 2020 Feb 24. PMID 32088984
- See also: PVDOMICS study protocol — http://lriapps.ccf.org/pvd/